CLINICAL TRIAL: NCT04923230
Title: Development of the Cannabis Actions and Practices (CAP): A Parent-Focused Intervention to Address Adolescent Marijuana Use
Brief Title: Pilot Test of Parent-Focused Cannabis-Related Actions and Practices Intervention for Adolescent Marijuana Abuse
Acronym: CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34DA049070 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-06-11 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cannabis Use Disorder, Mild; Cannabis Use Disorder, Moderate
Keywords: Adolescent; Marijuana Abuse; Prevention; Early Treatment
MeSH Terms: conditions — Lymphoma, Follicular; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: The pilot evaluation of CAP will be conducted with 60 MM parents who will be randomly assigned to CAP (n=30) or to a wait-list (WL) condition (n=30). Parents and their adolescents (n=120) will be assessed at baseline and at 3- and 6 months. WL parents will receive the CAP intervention after a 3-month waiting period and these participants will receive baseline and 3-month follow-up assessments. The study design and assessment schedule will allow both a between-groups test of the efficacy of CAP between intervention and delayed participants, as well as within-person test of pre- and post-intervention differences in the primary and secondary outcomes among all 60 parent/adolescent dyads.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors and investigators will not have knowledge of parent assignment to conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAP Intervention (Experimental): CAP is a parent-focused intervention being developed to help parents in states with legalized medical marijuana to address adolescent marijuana use. The proposed intervention will address the effects of marijuana on adolescent behavioral health, brain development, and social functioning and enhance parent motivation to use CAP concepts. Guided by formative research, CAP will build skills and provide strategies to: (1) restrict adolescent exposure to cannabis products and parent cannabis use in the home, (2) improve parent communication about their own cannabis use and expectations about youth marijuana use, (3) improve monitoring, (4) increase positive reinforcement for youth abstinence, and (5) address parent negative emotions. Parents will meet in groups with an interventionist for two 75-minute sessions. Presentations, discussion, and roleplay will be used to help parents gain mastery of preventive parenting behaviors and related strategies to reduce adolescent marijuana use.
  Interventions: Behavioral: Cannabis Actions and Practices Resource for Parents
- Wait List (No Intervention): Parents randomly assigned to Wait List Delayed CAP (WL) will receive no intervention for the baseline to 3-month follow-up period. Thus, the WL condition will serve as a comparison group from baseline to the 3-month assessment point. After the 3-month follow-up assessment, WL parents will be offered the CAP intervention. The final assessment for the WL participants will function as a 3-month follow-up assessment, allowing us to aggregate data all 60 parent-adolescent dyads to conduct within group analyses of pre- to post-intervention change on key variables of interest.

INTERVENTIONS:
Behavioral: Cannabis Actions and Practices Resource for Parents — The Cannabis Actions and Practices (CAP) resource is a parent-focused approach to help MM parents address marijuana use and attitudes by their adolescents. CAP includes information about the effects of marijuana on adolescent behavioral health, brain development, and social functioning. CAP also integrates motivational strategies to foster The CAP intervention focuses on building parenting skills and teaching strategies to: (1) limit adolescent exposure to cannabis products and parent cannabis use at home, (2) improve parent communication about their MM use, expectations about youth marijuana use, and attitudes about the potential harms of adolescent cannabis use, (3) improve monitoring, and (4) increase positive reinforcement for youth abstinence. Parents meet with an interventionist for two individual 75-minute sessions involving presentations, discussions, and behavioral rehearsal of key parenting skills.
  Other Names: CAP
  Arms: CAP Intervention

SUMMARY:
The randomized clinical trial involves the pilot-testing of a theory-guided, empirically based, and low-cost intervention designed for legal medical marijuana-using parents to enhance parenting behaviors that limit youth exposure to marijuana, reduce or halt youth marijuana use, and increase youth awareness of the harmful consequences of marijuana during the youth years. Parents will be randomized to an intervention condition or to a wait list control condition. Pre- and post-intervention assessments will evaluate parent and youth marijuana and other substance use, perceptions and attitudes about marijuana, parenting and family functioning, and youth behavioral health.

DETAILED DESCRIPTION:
The Stage 1A/1B treatment development research will involve a mixed-methods approach to formulating the Cannabis Actions and Practices (CAP) intervention. CAP is a parent-focused intervention to help parent medical marijuana (MM) users address adolescent marijuana use. The pilot evaluation of CAP will be conducted with 60 MM parents who will be randomly assigned to CAP (n=30) or to a delayed CAP wait-list (WL) condition (n=30). Parents and their adolescents will be assessed at baseline and 3, and 6 months after baseline. Primary outcomes will be adolescent marijuana use and perceptions of marijuana harmfulness. Secondary outcomes will include parenting behaviors such as youth exposure to marijuana, communications discouraging adolescent marijuana use, and setting expectations. The investigators will also examine key targets of change, including changes in adolescent behavioral health, parent perceptions of marijuana harmfulness, parent monitoring, parent sense of competence, parent behavioral intentions, and family relationships. Parents assigned to the delayed CAP condition will receive the CAP intervention after a 3-month waiting period, and these participants will receive baseline and 3-month follow-up assessments. The study design and assessment schedule will afford the opportunity for both a between-groups test of the efficacy of CAP between intervention and delayed participants, as well as within-person test of pre- and post-intervention differences in the primary and secondary outcomes among all 60 parent/adolescent dyads. The between-groups arm of the proposed design will provide an initial evaluation of the causal effects of the CAP intervention on primary and secondary marijuana use outcomes. The within-person arm of the design will provide an assessment of the degree to which participating parents improve in targeted areas of skill development and functioning after receiving the CAP intervention. All between-groups and within-person intervention effects will be evaluated within an intent-to-treat analytic framework. The study is designed to evaluate the promise of CAP, a novel theory-guided, empirically based, brief early intervention, for helping parent legal medical marijuana users support marijuana abstinence in their marijuana-involved adolescents.

ELIGIBILITY:
Parent Inclusion Criteria:

* Has a valid New Mexico medical marijuana card
* A biological or adoptive parent, step-parent or other parent figure who serves as the primary caregiver of a 13- to 17-year-old adolescent
* Parents and youth live together at least 40% of the time (i.e., minimum of 3 days per week)
* Reside in the greater Albuquerque, New Mexico area
* Has sufficient residential stability to permit probable contact at follow-up (e.g., not homeless at time of intake)
* Has sufficient English language skills to participate in the interventions and complete assessments

Adolescent inclusion criteria:

* Reports marijuana use on at least one occasion
* Has sufficient English language skills to complete assessments

Parent exclusion Criteria:

* Parent appears to have insufficient cognitive functioning to understand consent process, assessments and interventions
* Currently in drug treatment for a cannabis or other substance use disorder, whether medical or non-medical, and (3) a spouse or parenting partner is already enrolled in the study.

Adolescent exclusion criteria:

* Has a valid New Mexico medical marijuana card
* Reports weekly use of an illicit drug (i.e., excluding alcohol, tobacco, or marijuana)
* Appears to have insufficient cognitive functioning to understand assent process and assessments
* A sibling is already participating in the study

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adolescent Marijuana Use-Adolescent Report | baseline to 6-months
  The TLFB will be used to derive a measure of percent days of marijuana and other drug use in the past 12 weeks at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify change from baseline to 3-months and change from 3-months to 6-months.
Perceptions of Harmfulness of Marijuana Use Adolescent Report (PMHU-A) | baseline to 6-months
  The PMHU-A measure is based on items from the National Survey of Drug Use and Health (NSDUH). Five items from the NSDUH will be used to measure the respondent's perception about the harm of using marijuana pertaining to physical harm, harm to mental health, risk for marijuana dependence, risk for injuries, and harmful social consequences. Each item has the same response option (1=no risk, 2=some risk, 3=moderate risk, 4=high risk). Items will be summed to form a total score at each assessment point (range, 5-20), with the greater the scale score the more perceived risk. The PMHU will be used to derive a measure of perception of harm at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify change from baseline to 3-months and change from 3-months to 6-months.

SECONDARY OUTCOMES:
Cannabis-Specific Parenting Practices | baseline to 6-months
  The Cannabis-Specific Parent Practices measure will include: self-reported medical marijuana in the presence of youth, parents' verbal discouragement of youth marijuana use, parent-adolescent communication about parent expectations for abstinence, and parent safety protocols for cannabis storage at home. Parents will be asked to rate 7 items on a 4-point Likert-type scale (1= strongly disagree; 2=disagree; 3=agree; 4=strongly agree) regarding extent of agreement with each item. The greater the item score, the more optimal the parenting practice. Each item of this measure (score range, 1-4) will be collected at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed as separate items to quantify change from baseline to 3-months and change from 3-months to 6-months.

OTHER OUTCOMES:
Report of Parent Monitoring (PRM) Parent and Adolescent Forms | baseline to 6-months
  The Report of Parent Monitoring (PRM) will be used to measure parent level of involvement in and knowledge about their son's/daughter's social activities. The parent and adolescent versions of the scale each consists of 10 items (e.g., "I knew where my son/daughter was after school" and "my parents knew who friends were"), with responses ranging from "never or almost never" to "always or almost always" on a 5-point scale. Good internal consistency reliability and validity with alphas of .87 for reported. The greater the scale score (range, 10-50), the more optimal parental acceptance and involvement. Items will be summed for the parent and youth reports to form separate total PRM scale scores at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify parent and adolescent change from baseline to 3-months and change from 3-months to 6-months.
Family Environment Scale (FES)-Parent and Adolescent Forms | baseline to 6-months
  The Family Environment Scale (FES), a widely-used and well-standardized tool, is comprised of ten subscales which measure the quality of the family functioning. Moos and colleagues report internal consistency of the subscales ranging from .61 to .78, with test-retest reliabilities from .68 to .86 at 2-month intervals. The scale effectively distinguishes normal from disturbed families. The Conflict, Cohesion, and Organization subscales, key subscales for differentiating healthy and disturbed families and detecting pre-post treatment change, will be used. Each item has a True-False response option (1=true, 2=false), and the greater the scale score the more severe the family dysfunction. Items will be summed for parent and youth reports to form separate total FES scale scores at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify parent and youth change from baseline to 3-months and change from 3-months to 6-months.
Perceptions of Harmfulness of Marijuana Use-Parent Collateral Report (PHMU-P) and Self-Report (PHMU) | baseline to 6-months
  The PHMU-P is based on items from the National Survey of Drug Use and Health (NSDUH). The 5-item PHMU-A will be modified to ask parents about the level of risk of marijuana use for teenagers. Risk scores will be summed to form a total score. Parents will also be asked to respond to the 5 PHMU items pertaining to their perception of risk of their own marijuana use to aid in characterizing the study sample. Each item for PHMU-P and PHMU has the same response option (1=no risk, 2=some risk, 3=moderate risk, 4=high risk). Items will be summed to form a total score at each assessment point for each scale (range, 5-20), with the greater the scale score the more perceived risk. The PMHU-P and PMHU will be used to derive separate measures of perception of harm at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify change from baseline to 3-months and change from 3-months to 6-months.
Behavioral Intentions Questionnaire (BIQ) Parent Report | baseline to 6-months
  The Behavioral Intentions Questionnaire (BIQ) is a 6-item scale designed to assess parent likelihood of applying the intervention concepts, strategies, and skills in their home environment. Behavioral intentions and expectations assess an individual's perceived likelihood of future behavior. BIQ items include parent intentions to restrict adolescent exposure to cannabis at home and parent intentions to provide messages to their adolescent that discourage underage use. Responses will be rated on 4-point Likert type scale ranging from "very likely" to "very unlikely". Ratings will be summed to provide a total BIQ score (range=6-24). The greater the scale score, the greater the perceived intention to use the resource. The BIQ will be used to derive a measure of likelihood to use the resource in the future at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify change from baseline to 3-months and change from 3-months to 6-months.
Parent Sense of Competence Scale (PSOC) Parent Form | baseline to 6-months
  Parent efficacy and satisfaction in their own parenting will be assessed with the Parent Sense of Competence scale (PSOC), a 17-item questionnaire with items on a 4-point scale (1=strongly agree, 2=agree, 3=disagree, 4=strongly disagree). The subscales have adequate internal consistency (alpha=.82 for Satisfaction, alpha =.70 for Efficacy). Satisfactory test-retest correlations for the scales and total score were also reported. Items will be added to the PSOC to assess parents' perceptions of their self-efficacy with respect to performing the strategies and skills presented in the intervention. Ratings will be summed to provide a total PSOC score (range=17-68). The greater the scale score, the greater the perceived parenting efficacy. The PSCO will be used to derive a measure of perceived parenting at three time points (baseline, 3-months follow-up, and 6-months follow-up) and analyzed to quantify change from baseline to 3-months and change from 3-months to 6-months.
Urine Toxicology Screen-Parent | baseline to 6-months
  Urine toxicology screening will be conducted to verify parent report of substance use. Recent drug use will be measured using Urine Assays (UA; NIDA 12 Test Panel), using a card device with 12 finger-like prongs dipped in a urine sample will screen youth for amphetamine, barbiturates, benzodiazepines, cocaine, ecstasy, meth-amphetamine, methadone, opiates, oxycodone, phencyclidine, tricyclics, and marijuana, plus three adulterants, providing a verification of self-report. Test cups will monitor temperature to further detect tampering. Clear results for photocopy emerge within 5 minutes to simplify data collection by trained project staff. All samples will be discarded once the results have been documented. UAs, consequences and other substance use variables will be used to aid with the interpretation of study findings. Urine screen results at each time point will be compared to substance use self-report at the respective time point.
Parent Cannabis Use (DFAQ-CU) | baseline, to 6-months
  Parent cannabis use quantity and frequency will be measured using the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis-Use Inventory (DFAQ-CU; Cuttler & Spradlin, 2017). The DFAQ-CU shows pictures of various marijuana quantities to assess the quantity of cannabis used for various forms of cannabis, different methods of administration, amounts used, and typical THC levels in cannabis used. The DFAQ-CU has favorable internal reliability for the 6 factors (alpha range, .69 to .95) and favorable evidence for convergent, predictive, and discriminant validity. The range of scale scores vary across subscales, yet for each the greater the subscale score, the more use of marijuana is indicated. Subscale scores will be summed to form a total score at each time point (baseline, 3-months follow-up, and 6-months follow-up) and quantify change from baseline to 3-months and change from 3-months to 6-months.
Timeline Follow-back (TLFB) Parent Report | baseline to 6-months
  Timeline Follow-back Interview (TLFB) will also be used to measure the parents past 12 weeks of use of other licit and illicit substances and of nonmedical and medical marijuana use. This instrument is a structured interview that yields a daily calendar-aided reconstruction of use from all drug classes (including alcohol) to facilitate recall and minimize retrospective biases. TLFB is sensitive treatment-related change, has good psychometric properties, and produces higher estimates of use than summary measures. Direct self-report measures compare favorably to collateral reports and have been validated using urine toxicology screening. Parent substance use data at baseline will be used for sample characterization and to guide interpretation of study findings (change across time).
Adolescent Strengths and Difficulties Questionnaire (SDQ) Parent Report | baseline
  The Strengths and Difficulties Questionnaire (SDQ) (Goodman, 1997) will be used to measure the parent's perception of youth difficulties and prosocial competence. The SDQ is an internationally-validated 25-item questionnaire comprised of five subscales: emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior. Each item is responded to on a 3-point ordinal scale, ranging from 0 = not true to 2 = certainly true. Subscale scores range from 0-10, and the total SDQ score ranges from 0 to 40, with higher scores indicating more problems and less competence. The SDQ has high discriminant validity and is predictive of child internalizing and externalizing behavior (Goodman, 1997; Goodman & Scott, 1999). SDQ scales at baseline will be used to characterize the study sample.

CONTACTS AND LOCATIONS:
Overall Officials: Holly B Waldron, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Center for Family and Adolescent Research, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available 5 months after publication of initial study findings and will be available for a period of 2 years.
Access Criteria: Data will be shared with behavioral health researchers by written request for further analysis and publication of findings. The MPIs for the study will review requests. Review criteria to be determined.